CLINICAL TRIAL: NCT01165047
Title: An Open Label, Non-Randomized Pilot Study to Evaluate the Safety and Performance of the GeNO Nitrosyl Delivery System in Subjects Being Evaluated for Orthotopic Heart Transplantation (OHT), or Left Ventricular Assist Device (LVAD) Implantation
Brief Title: Nitric Oxide, GeNO Nitrosyl Delivery System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2014-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitric Oxide (Experimental): 80 ppm in air or oxygen will be administered using the GeNO nitrosyl delivery system with a standard nasal cannula at a flow rate of 4 LPM
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Nitric oxide, 80 ppm in air or oxygen will be administered using the GeNO nitrosyl delivery system with a standard nasal cannula at a flow rate of 4 LPM.
  Other Names: GeNO nitrosyl delivery system

SUMMARY:
The primary aim of the study is to evaluate the safety, tolerability and device performance of the GeNO nitrosyl delivery system during RHC. Secondary considerations are to confirm that inhaled NO generated by the GeNO nitrosyl delivery system, reduces PVR in patients with reversible PH, contains levels of NO2 well below the upper level of acceptable exposure. Further, the study aims to demonstrate that patient response to inhaled NO can be used as a diagnostic tool with which to determine the proper course of medical action in patients with chronic heart failure.

Patients with chronic heart failure accompanied by pulmonary hypertension and increased pulmonary vascular resistance have a number of possible medical therapies available to them. The least invasive, and therefore most appealing, option is standard management with medication and observation. Alternatively, implantation of a left ventricular assist device (LVAD) may be considered, either as a permanent solution or as a bridging strategy to the final option, orthotopic heart transplantation (OHT). It is often unclear which route is the best medical choice, and a tool to help physicians and patients choose between these alternatives would be greatly beneficial.

It has been shown that chronic heart failure patients that demonstrate irreversible pulmonary hypertension, even in the presence of vasodilators, exhibit adverse outcomes after OHT (Tsai et al., 2002; Ericson et al., 1990; Murali et al., 1996). It follows that patient response to pulmonary vasodilators can, and should be used to classify patients as potential candidates for OHT. In particular, patient response to inhaled NO, a known pulmonary vasodilator, can be used as a diagnostic tool to assist in deciding which medical route to take.

With this in mind, the current study aims to demonstrate whether or not NO generated by the GeNO nitrosyl delivery system effects a reduction in pulmonary hypertension due to increased pulmonary vascular resistance in patients with chronic heart failure. Any demonstrated ability of inhaled NO to decrease PVR in patients with reversible PH will support the use of patient response to inhaled NO as a diagnostic tool to assist in choosing the most appropriate medical therapy for patients with chronic heart failure.

DETAILED DESCRIPTION:
Investigational product will be administered by qualified study staff in accordance with the procedures described in the protocol and in accordance with the detailed set of instructions supplied with the initial shipment of investigational product.

Nitric oxide, 80 ppm in air or oxygen will be administered using the GeNO nitrosyl delivery system with a standard nasal cannula at a flow rate of 4 LPM.

In order to reliably measure trace levels of NO2 in the presence of a large excess of NO, it is essential to use a technique with extremely high accuracy in situations of low levels of NO2. The GeNO nitrosyl delivery system delivers a fixed concentration of 80ppm NO with low levels of NO2 which current technology cannot measure with accuracy at levels below 3ppm.

The investigational product is the GeNO nitrosyl delivery system which consists of a drug/device combination product with all the components necessary to deliver the investigational drug; the nitric oxide gas. The investigational drug, nitric oxide, is generated at the time of use when the NO2 input gas flows through the cartridge, the antioxidant reduces the NO2 to NO.

The input gas is supplied as either nitric oxide in air or nitric oxide in oxygen. The Investigator will determine whether air or oxygen is used as the balance gas, on the basis of the participant's clinical needs for supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review board (IRB) approved informed consent is signed, dated and timed prior to any study-related activities.
* Male or female > 18 years of age.
* Being evaluated for OHT or LVAD implantation and scheduled to undergo right heart catheterization to assess pulmonary vasoreactivity.
* Have a confirmed diagnosis of heart failure, (NYHA Class III or IV)
* Participant has the ability to understand the requirements of the study and a willingness to comply with all study procedures.
* Females of childbearing potential with a negative urine pregnancy test, or a documented surgical sterilization, or is post-menopausal prior to administration of investigational product. Females of childbearing potential must be practicing adequate birth control to be eligible. It is the Investigator's responsibility to determine whether the Participant has adequate birth control for study participation.
* Confirmed pulmonary arterial hypertension at time of RHC:

  * PAPm > 25mmHg at rest and PVR > 3 Wood units

Exclusion Criteria:

* Be receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within the past 30 days.
* Have had an atrial septostomy.
* Have anemia (hemoglobin <10 g/dL), active infection or any other ongoing condition that would interfere with the interpretation of study assessments.
* Have any serious or life-threatening disease other than conditions (e.g. malignancy requiring aggressive chemotherapy, etc.).
* Have unstable psychiatric status or be mentally incapable of understanding the objectives, nature or consequences of the trial, or any condition, which in the investigator's opinion would constitute an unacceptable risk to the participant's safety.
* Participant is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Boyle, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitric Oxide
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nitric Oxide
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants] — >= 18 years
  participants
    equal or greater than 18 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Effects and/or Adverse Events
Description: A phone contact will be made to the subject 5 days after the trial to assess general health status and collect information on any reported side effects or adverse events.
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Nitric Oxide
Number analyzed (Participants) | 8
participants | 0

ADVERSE EVENTS:
Arm/Group | Nitric Oxide
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No